CLINICAL TRIAL: NCT01170338
Title: Safety and Efficacy of the Novel Selective Nicotinic Receptor Partial Agonist, CHANTIX (Varenicline) in Patients With Acute Coronary Syndrome
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Newark Beth Israel Medical Center (Other)
Responsible Party: Marc Cohen, MD, Newark Beth Israel Medical Ctr
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2008.68
Record Dates: First submitted 2010-07-26; First posted 2010-07-27 (Estimated); Last update posted 2010-07-27 (Estimated); Status verified 2010-07

CONDITIONS: Smoking; Acute Coronary Syndrome
Keywords: smoking; tobacco abuse
MeSH Terms: conditions — Smoking; Acute Coronary Syndrome; Tobacco Use Disorder | interventions — Varenicline

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- active Chantix (Experimental): active drug to help smoking cessation
  Interventions: Drug: Varenicline 100 mg by mouth twice daily
- sugar pill (Placebo Comparator)
  Interventions: Drug: control

INTERVENTIONS:
Drug: Varenicline 100 mg by mouth twice daily — this is an active drug to help smoking cessation
  Arms: active Chantix
Drug: control — this is the placebo that will help us maintain a blinded study
  Arms: sugar pill

SUMMARY:
Assess the role of a nicotine antagonist in helping patients presenting to hospital with acute coronary syndrome to stop smoking.

ELIGIBILITY:
Inclusion Criteria:

* active smokers presenting to hospital with an acute coronary syndrome

Exclusion Criteria:

* patients with an acute coronary syndrome who are not active smokers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2008-01; Primary Completion 2011-07 (Estimated)

PRIMARY OUTCOMES:
nicotine levels | 1 month

SECONDARY OUTCOMES:
recurrent myocardial ischemia | 1 month

CONTACTS AND LOCATIONS:
Locations (1):
- Newark Beth Israel Medical Center, Newark, New Jersey, United States